CLINICAL TRIAL: NCT04633577
Title: The Effect of Intravenous Lidocaine on Propofol Requirements in Patients Undergoing Hysteroscopy and Diagnostic Curettage
Brief Title: Effect of Intravenous Lidocaine on Propofol Requirements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020-1000
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2020-11

CONDITIONS: Analgesia
Keywords: intravenous lidocaine; propofol; pain score; fatigue score; dose
MeSH Terms: conditions — Agnosia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Lidocaine (Experimental): 20 eligible patients are received 1.5mg/kg 1%lidocaine intravenously over 30-60s. Then, 4mg/kg/h lidocaine infused intravenously until end of procedure.
  Interventions: Drug: Lidocaine IV
- Group Control (Placebo Comparator): 2020 eligible patients are received equal 0.9% normal saline.
  Interventions: Drug: 0.9% normal saline

INTERVENTIONS:
Drug: Lidocaine IV — A bolos of 1.5mg/kg lidocaine will be administered before induction. Then, infusion of 4mg/kg/h lidocaine will maintain during procedure.
  Arms: Group Lidocaine
Drug: 0.9% normal saline — 0.9% normal saline
  Arms: Group Control

SUMMARY:
Lidocaine, an amide local anesthetic, has advantages of low price and easily obtaining. Intravenous lidocaine (IVL)initially has been used in the treatment of arrhythmia. It was demonstrated that IVL had analgesic effect, especially in colorectal surgery, but remained controversy in other types of surgeries. Other beneficial effects, such as prevention of hyperalgesia and propofol-induced injection pain, reduction of incidence of postoperative ileus and nausea and vomiting and anti-inflammatory also were proposed.

DETAILED DESCRIPTION:
The most frequent drugs for procedural sedation and analgesia are propofol, benzodiazepines and opioids. However, these drugs may cause respiratory depression and circulatory instability. Combination will increase the risk of hypoxia and apnea.

In China, most anesthesia for hysteroscopy and gastroenteroscopy is procedural sedation and analgesia(PAS) provided by anesthetists. Foester et,al. have been tested that IVL could significantly reduce propofol requirements 、postoperative pain and fatigue scores in colonoscopy. Chen,et,al. find the same effect of IVL in elderly. However, there is no research reporting IVL used in hysteroscopy and diagnostic curettage. So, our main objective is to evaluate the effect of intravenous lidocaine on propofol requirements in patients undergoing hysteroscopy and diagnostic curettage.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent hysteroscopy and diagnostic curettage, American Society of Anesthesiologist' physical status 1-2, BMI 18.5-24.9 kg/m2,

Exclusion Criteria:

* Patients with known allergy to lidocaine or other local anesthetics, taken sedatives and analgesics within 1 week before surgery, mental and neurological diseases, hearing impairment, unwilling to sign informed consent or participate in the study, serious arrhythmia and organic heart disease.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female could undergo hysteroscopy and diagnostic curettage
Enrollment: 40 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Propofol Requirements | from loss of conciousness to end of procedure
  propofol requirements at loss of conciousness and supplemental requirements during procedure

SECONDARY OUTCOMES:
Pain score | immediately, 15 min, 30 min in PACU
  Assessed pain score using 0-10 cm VAS
Fatigue score | immediately, 15 min, 30 min in PACU
  Assessed fatigue score using 0-10 cm VAS

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

REFERENCES:
- [Background] Forster C, Vanhaudenhuyse A, Gast P, Louis E, Hick G, Brichant JF, Joris J. Intravenous infusion of lidocaine significantly reduces propofol dose for colonoscopy: a randomised placebo-controlled study. Br J Anaesth. 2018 Nov;121(5):1059-1064. doi: 10.1016/j.bja.2018.06.019. Epub 2018 Aug 1. PMID 30336850
- [Background] Chen M, Lu Y, Liu H, Fu Q, Li J, Wu J, Shangguan W. The propofol-sparing effect of intravenous lidocaine in elderly patients undergoing colonoscopy: a randomized, double-blinded, controlled study. BMC Anesthesiol. 2020 May 30;20(1):132. doi: 10.1186/s12871-020-01049-z. PMID 32473649